CLINICAL TRIAL: NCT02262949
Title: A Prospective Study of the Bard® LifeStent® Solo Vascular Stent System (REALITY2)
Brief Title: A Prospective Study of the Bard® LifeStent® Solo Vascular Stent System
Acronym: REALITY2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-13-002; DRKS00006281 (Registry Identifier: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2014-09-25; First posted 2014-10-13 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LifeStent Vascular Stent (Experimental): This is a single arm study and all subjects receive PTA and implantation of one Life Stent Vascular Stent.
  Interventions: Device: LifeStent Vascular Stent

INTERVENTIONS:
Device: LifeStent Vascular Stent — PTA followed by implantation of the LifeStent Vascular Stent (stent length 250 mm) in the SFA or popliteal artery.

SUMMARY:
The purpose of this study is to assess the deliverability, clinical utility, safety and effectiveness of the 250 mm length size offering of the LifeStent® Vascular Stent.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legal representative has been informed of the nature of the evaluation, agrees to its provisions, and has signed the informed consent form (ICF).
2. Subject agrees to comply with the protocol-mandated follow-up procedures and visits.
3. The subject is ≥ 21 years old.
4. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within seven days prior to index procedure. Female subjects who are surgically sterile or post-menopausal are exempt from having a pregnancy test.
5. The subject has lifestyle-limiting claudication or mild tissue loss defined as: Rutherford Category1 2-5 (moderate claudication to minor tissue loss).
6. The target lesion has angiographic evidence of stenosis or restenosis ≥50% or occlusion in the SFA and/or popliteal artery (by visual estimate) and is amenable to PTA and stenting.
7. The target vessel reference diameter is (by visual estimate) appropriate for treatment with available stent diameters of 6.0 and 7.0 mm.
8. There is angiographic evidence of at least one vessel runoff to the foot (at the level of the malleolus).

Exclusion Criteria:

1. The subject is unable or unwilling to provide informed consent or is unable or unwilling to comply with the study follow-up procedure and visits.
2. The subject has claudication or critical limb ischemia described as Rutherford Category 0 (asymptomatic), 1 (mild claudication), or 6 (major tissue loss).
3. The subject has a known contraindication (including allergic reaction) or sensitivity to antiplatelet/anticoagulant medication, nickel, titanium or tantalum.
4. The subject has a known sensitivity to contrast media that is not amenable to pretreatment with steroids or/and antihistamines.
5. The subject has a history of bleeding diatheses of coagulopathy.
6. The subject has concomitant renal failure with a creatinine of >2.5 mg/dL.
7. The subject has concomitant hepatic insufficiency,thrombophlebitis, uremia, systemic lupus erythematosus (SLE), or deep vein thrombosis (DVT) at the time of the study procedure.
8. The subject is receiving dialysis or immunosuppressive therapy.
9. The subject is participating in an investigational drug or another investigational device study.
10. The subject has another medical condition, which, in the opinion of the investigator, may cause him/her to be noncompliant with the protocol, confound the data interpretation, or is associated with limited life expectancy of less than two years.
11. The subject has extensive peripheral vascular disease, which,in the opinion of the investigator, precludes safe insertion of an introducer sheath.
12. The target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion.
13. The subject has angiographic evidence of poor inflow, which would be deemed inadequate to support a vascular bypass graft.
14. The subject is diagnosed with septicemia at the time of the study procedure.
15. Subjects with a stent previously implanted into the target lesion. A target vessel with a previously placed stent is permitted as long as the subject device will not come into contact with the previously placed stent during treatment of the target lesion.
16. Lesions requiring the use of more than one investigational stent.
17. Bilateral disease in the native SFA and/or proximal popliteal artery where both limbs meet the inclusion/exclusion criteria and it is planned to treat both limbs within 30 days.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events (MAEs) | 30 days
  Occurence of death or target limb amputation or any target lesion revascularization/target vessel revascularization through 30 days post-index procedure. These events will be assessed by clinical evaluations.
Stent performance | intra operative
  Stent deployment success; defined as a post-deployment stent length deviating <10% from pre-deployment stent length (determined by an independent core lab).
  Placement accuracy based upon a rating scale completed by the investigator at time of index procedure.

SECONDARY OUTCOMES:
Major Adverse Events (MAEs) | 1 year
  Occurence of death, stroke, MI, emergent surgical revascularization of the target limb, significant distal embolization in target limb, target limb major amputation, and thrombosis of target vessel at 12 months post-index procedure. These events will be assessed by clinical evaluations.
Target lesion/vessel revascularization | 1 year
  TLR/TVR rate after 12 months post-index procedure. TLR/TVR will be assessed by clinical evaluations.
Target lesion patency | 1 year
  Primary patency (PSVR<2.4) rate at 12 month post-index procedure (measured by DUS). Patency will be assessed by clinical evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof. Dr., Principal Investigator — University Heart Centre Freiburg, Bad Krozingen
Locations (4):
- Germany (4):
  - University Heart Centre Freiburg, Bad Krozingen
  - Gemeinschaftspraxis für Radiologie, Berlin
  - Fürst Stirum Klinik Bruchsal, Bruchsal
  - RoMed Klinikum Rosenheim, Rosenheim